CLINICAL TRIAL: NCT02862249
Title: A Prospective, Randomised Placebo Controlled Feasibility Trial of Faecal Microbiota Transplantation in Cirrhosis
Brief Title: Trial of Faecal Microbiota Transplantation in Cirrhosis
Acronym: PROFIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PROFIT-01
Record Dates: First submitted 2016-02-05; First posted 2016-08-11 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cirrhosis of the Liver
MeSH Terms: conditions — Fibrosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faecal microbiota transplantation (Experimental): Faecal microbiota transplantation.
  Interventions: Biological: Faecal microbiota transplantation
- Placebo (Placebo Comparator): Placebo solution.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Faecal microbiota transplantation — The FMT (200mls) will be administered following preparation of the bowel with MoviPrep®, into the duodenum via a gastroscope derived from 50g of fresh donated stool from a healthy donor. The gastroscopy will be performed as per the King's College Hospital Gastroenterology Protocol.
  Arms: Faecal microbiota transplantation
Biological: Placebo — An identical appearing placebo solution (200mls 0.9% normal saline and 12.5% glycerol) will be administered into the duodenum via a gastroscope in a single blinded fashion following preparation of the bowel with MoviPrep®.
  Arms: Placebo

SUMMARY:
Patients with advanced cirrhosis have enteric dysbiosis with small bowel bacterial overgrowth and translocation of bacteria and their products across the gut epithelial barrier. This culminates in systemic inflammation and endotoxemia which induces innate immune dysfunction predisposing to infection and development of complications such as bleeding, sepsis and hepatic encephalopathy. It also plays a key role in the natural history of cirrhosis by influencing the rate of progression to advanced liver disease and terminal liver failure.

The investigators propose an intervention utilising Faecal Microbiota Transplantation (FMT) from a healthy donor to modify the gut microbiome alleviating gut dysbiosis and immune dysfunction. This may ultimately reduce the progression to chronic liver failure and the development of infection and organ dysfunction.

The primary objective of this study will be to assess whether stabilising gut dysbiosis with FMT in patients with advanced cirrhosis is both feasible and safe.

DETAILED DESCRIPTION:
Humans are colonized by a diverse range of microbes, the most abundantly inhabited being the gastrointestinal tract which anatomically commences at the oral mucosa, with the colonic lumen being the most densely populated. The gut microbiota consist mainly of bacteria, but it is worth remembering that fungi, viruses, archaea and protozoa are also resident and active. As a composite, these micro-organisms outnumber human cells by a factor of ten. Humans can carry up to two kilograms of microbes within our gut, and these tens of trillions of micro-organisms have been referred to as the 'last human organ.' Whilst these microbes consist of over three million genes, or an impressive 150 times the number contained within our own genome, two thirds of the entire gut microbiome is unique to each individual. Furthermore although the gut microbiome consists of greater than 1,000 species of bacteria; approximately 170 species predominate in any given individual with Bacteroidetes and Firmicutes being the dominant phyla. The diverse and complex role played by the gut microbiome includes the development and modulation of the innate and adaptive immune systems; both locally within the intestinal mucosa with defense against pathogens and tumorigenesis, and systemically. Dietary and homeostatic functions pertain to the biosynthesis of vitamins, metabolism of glucose, bile salts and xyloglucans, and the liberation of short-chain fatty acids (SCFAs) from otherwise indigestible dietary starches, mainly by bacteria from the Bacteroidetes phylum. SCFAs have immune-signaling and anti-inflammatory properties and are a vital source of energy for intestinal mucosal cells helping to maintain intestinal integrity and barrier function. A change to the gut microbiome therefore impacts on a multitude of vital homeostatic functions, many of which the human host cannot perform independently.

Technological advances in genomic sequencing and bioanalytics are beginning to revolutionize our understanding of the gut microbiome in relation to hepatological diseases. Further insights are now being gained with the unraveling of some of the complex mechanisms that contribute to the commensal and synergistic interactions between the host and our microbiome, and the downstream mechanistic effects in both normal physiology and when these processes are disturbed inducing pathology. It is well established that patients with cirrhosis have enteric dysbiosis with small bowel bacterial overgrowth and translocation of bacteria and their products (such as lipopolysaccharide and bacterial DNA) across a more permeable gut epithelial barrier which is exacerbated by underlying portal hypertension and endothelial dysfunction. This culminates in systemic inflammation and endotoxemia which induces innate immune dysfunction via toll-like receptor signaling, predisposing to infection and development of decompensating complications such as haemorrhage, sepsis and hepatic encephalopathy (HE). Indeed, it is widely recognised that intestinal decontamination with non-absorbable antibiotics such as rifaximin is an effective treatment for HE. This implicates gut dysbiosis and the ensuing metabolic sequelae involving intestinal absorption of nitrogenous compounds in the progression of neurocognitive dysfunction.

Enteric dysbiosis has also been linked to progression to advanced liver disease. Utilising quantitative metagenomics it has been recently shown that 75,245 microbial genes differ in abundance between patients with cirrhosis and healthy individuals, and of relevance that over 50% of these taxonomically assigned bacterial species are of buccal origin suggesting an invasion of the gut from the mouth in cirrhosis. Salivary dysbiosis, represented by a reduction in autochthonous bacteria, is also present and to an extent reflects the changes seen in the faecal microbiota in cirrhosis, with an associated systemic and salivary-specific inflammatory milieu.

Of note salivary dysbiosis is more pronounced in patients that go on to be hospitalized during 90-day followup.

This implies a causative role particularly when considering that cirrhotic saliva is enriched with genes related to endotoxin synthesis proteins, and nucleic acid and vitamin metabolism, the latter of which are purported to modulate intestinal barrier integrity and oxidative stress. Modulating the gut microbiota in patients with cirrhosis with the non-absorbable antibiotic rifaximin has been associated with improved cognitive performance and reduction in endotoxemia in patients with cirrhosis.

Moreover, the investigators have recently performed a multicentre retrospective study including 170 patients in which rifaximin therapy given for 90-days significantly (i) reduced hospital re-admission rates after 3 months treatment, impacting significantly on the NHS resource burden and (ii) reduced overall liver disease severity [as measured by the Child Pugh and Model for End Stage Liver Disease scores raising the possibility that modulation of gut microbiota may significantly modify the natural history of chronic liver failure.

These data constitute in the investigators' view "proof of principle" that modifying the gut microbiota in patients with cirrhosis improves clinical outcomes. Rifaximin was approved by NICE for the prevention of the recurrence of overt hepatic encephalopathy in cirrhosis, but considerable concern remains regarding whether long term antibiotic prescription will result in a change in bacterial function and virulence rather than a simple reduction in bacterial population and whether this may drive bacterial resistance to antibiotics in an already functional immunocompromised population. The question therefore is raised as to whether directly, as opposed to indirectly modulating the gut microbiota utilising faeces from healthy donors may be a safer and more durable therapy. Faecal microbiota transplantation (FMT) is a well-established treatment to stably modify the gut microbiome and has been shown to be safe and efficacious in several disease states resulting from gut dysbiosis including Clostrium difficile infection [NICE approved] and inflammatory bowel disease.

The investigators hypothesize that in patients with advanced cirrhosis FMT may reduce the progression to chronic liver failure including jaundice, accumulation of fluid within the abdominal cavity, bleeding, encephalopathy and the development of infection and organ dysfunction. Whether FMT is feasible in the setting of liver cirrhosis remains to be investigated. A trial is proposed to determine whether a FMT from a healthy donor to a patient with advanced cirrhosis is both feasible and safe.

ELIGIBILITY:
Inclusion criteria:

* 18-75 years
* Confirmed advanced cirrhosis of any aetiology with a MELD score between 10 and 16. The diagnosis of liver cirrhosis will be based on clinical, radiological, or histological criteria.
* Patients with alcohol-related liver disease must have been abstinent from alcohol for a minimum of 6 weeks.
* Patients must be deemed to have capacity to consent to study.

Exclusion criteria:

* Severe or life-threatening food allergy
* Pregnancy or breastfeeding
* Patients treated for active variceal bleeding, infection, bacterial peritonitis, overt hepatic encephalopathy or acute-on-chronic liver failure within the past 14 days.
* Patients who have received antibiotics in the past 14 days.
* Active alcohol consumption of >20 grams/day.
* Has had a previous liver transplant
* Hepatocellular carcinoma outside of the Milan Criteria (2)
* A history of prior gastrointestinal resection such as gastric bypass
* Patient is not expected to survive the duration of the study (90 days).
* Severe renal impairment (creatinine >150 µmol/L)
* Inflammatory bowel disease (IBD)
* Coeliac disease
* HIV positive
* Immunosuppression e.g. more than two weeks treatment with corticosteroids within 8 weeks of intervention, active treatment with tacrolimus, mycophenylate, azathioprine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Assessment of the feasibility of FMT | 18 months
  Assess recruitment rates and tolerability of FMT (e.g reflux rates):
  * >50% fulfil inclusion/exclusion criteria (of all screened- about 160)
  * >25% consent rate (of all those fulfilling inclusion/exclusion criteria about 80 patients)
  * >80% randomised patients treated successfully and completing study up to D90 (out of those randomised approx 22 patients)
  * Availability of obtaining sufficient donor samples for the study
  * Reflux rates of transplanted material <20% e.g. foul taste, foul smell, nausea, vomiting, indigestion.
  * Intolerable (resulting in withdrawal from the study GI side effects including diarrhoea, constipation, abdominal pain, flatulence and bloating) of <20%
Assessment of the Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 18 months
  1. Incidence of any transmissible bacterial or viral infection that is deemed to have been acquired from the donor including Clostridium Difficile infection
  2. The development of any SAE/SAR or USAR that is not pre-specified or is a known consequence of disease progression or complication of cirrhosis as outlined in section 7.2.5.1 that: results in death/is life threatening/requires hospitalisation or prolongation of existing hospitalisation/results in persistent or significant disability or incapacity.

SECONDARY OUTCOMES:
To provide preliminary evidence of efficacy for a larger randomised trial | 18 months
  (i) Choosing the optimal primary outcome, and (ii) Estimating the parameters for sample size calculation.
To estimate the costs and resources required to implement this novel therapy in a NHS environment. | 18 months
  Cost effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Shawcross, Study Chair — King's College London
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All information, data and results obtained from study are confidential. Agreement from the Sponsor will be required prior to the public disclosure of any study-related data. It is expected that results from the study will be published in peer-reviewed scientific/medical journals and presented at scientific/clinical symposia and congresses. All publications and presentations relating to the study must be authorised by the CI.

REFERENCES:
- [Derived] Woodhouse CA, Patel VC, Goldenberg S, Sanchez-Fueyo A, China L, O'Brien A, Flach C, Douiri A, Shawcross D. PROFIT, a PROspective, randomised placebo controlled feasibility trial of Faecal mIcrobiota Transplantation in cirrhosis: study protocol for a single-blinded trial. BMJ Open. 2019 Feb 15;9(2):e023518. doi: 10.1136/bmjopen-2018-023518. PMID 30772848